CLINICAL TRIAL: NCT01437280
Title: GOAT; Phase I Single-Center Open Label Dose Escalation Study of CGTG-102, a GM-CSF Encoding Oncolytic Adenovirus, for Therapy of Advanced Cancers
Brief Title: GOAT; Phase I Open Label Study of CGTG-102, a GM-CSF Encoding Oncolytic Adenovirus, for Advanced Cancers
Acronym: GOAT
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: The Methodist Hospital Research Institute (Other); Harris County Hospital District (Other Government)
Responsible Party: Principal Investigator, Martha Mims, Principal Investigator, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-28686-GOAT; GOAT (Other: CAGT/BCM)
Record Dates: First submitted 2011-09-15; First posted 2011-09-20 (Estimated); Last update posted 2013-08-14 (Estimated); Status verified 2013-08

CONDITIONS: Tumors; Solid Tumors
Keywords: Tumors; Solid Tumors
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CGTG-102 (Experimental): CGTG-102 is an oncolytic adenovirus
  Interventions: Biological: CGTG-102

INTERVENTIONS:
Biological: CGTG-102 — VP=virus particle
  Dose Level 1: 3x10^10 VP/injection
  Dose Level 2: 1x10^11 VP/injection
  Dose Level 3: 3x10^11 VP/injection
  Patients will receive 4 administrations of CGTG-102 (on days 1, 4, 8, 15).
  Escalation to the next dose level will occur when the safety of all 4 administrations has been evaluated at day 43 on all patients in the preceding dose level.
  The total dose will be injected into up to 10 tumors injectable by either direct visualization/palpitation and/or ultrasound. Typically, the largest safely injectable tumors are chosen.
  Injections will be performed by a radiologist or other trained physician. Injections will be planned based on the baseline PET-CT: only PET-positive tumors or tumor regions should be injected. Injection needles designed for percutaneous insertion into tissues will be used.

SUMMARY:
Oncolytic viruses are viruses that can be found in nature, but they have been modified so that they can no longer multiply in normal cells. These viruses "infect" cancer cells and kill them. Once the cancer cell dies thousands of the viruses are released and can potentially infect other cancer cells in the area. The effects of oncolytic viruses on the tumor are felt to be the result of a combination of the oncolytic viruses directly killing the tumor cells as well as the patient's immune system killing cancer cells that are infected with the oncolytic virus.

Modern oncolytic viruses have been used for treatment of thousands of patients. The safety of such treatments has been good and there have been no deaths caused by treatment with oncolytic viruses. Many patients have benefited from the treatment in the sense that their tumors have stopped growing, become smaller or even completely disappeared. Some benefits are temporary, but about one third of patients seem to gain longer lasting benefit likely to impact survival. The effect of oncolytic viruses on improving survival has not been demonstrated yet.

Oncolytic viruses can be created from many different types of viruses. In this study the investigators are using an oncolytic virus created from an adenovirus. Adenoviruses are the types of viruses that cause the common cold and the flu. Because replication in normal cells does not take place, these oncolytic viruses should not cause any diseases in normal cells. Further, to date there has been no incidence of passing the virus on to other humans from patients who were treated with oncolytic viruses.

The purpose of this study is to see the highest dose of CGTG-102 (the oncolytic virus being used in this study) that can safely be given to subjects. The investigators will also evaluate whether or not the CGTG-102 is helpful in reducing the size of the cancer and improving patient survival.

DETAILED DESCRIPTION:
Pre-treatment visit - subject will undergo a physical examination with vital signs, a blood sample will be taken and a PET (Positron emission tomography)-CT (Computer tomography) scan will be performed.

Thereafter, there will be 4 visits with injections performed on trial days 1, 4, 8 and 15.

TREATMENT:

The injections are given directly into the tumors with help from using an ultrasound. The total dose of oncolytic virus the subject will receive will be divided into 1-10 injections which will be injected into individual tumors in the body. The maximum number of tumors that can be injected for one treatment will be 10 tumors.

STUDY VISIT 1:

On the day 1 visit, blood samples will be taken as well as two biopsies from one of the tumors. In addition pleural fluids (fluids from the chest) or ascites (fluids from abdominal walls) may be collected if possible. Then the subject will receive the first set of injections with CGTG-102. Before the injections, the subject may be given a dose of Tylenol.

STUDY VISIT 2:

On the day 4 visit, in addition to blood samples being taken the subject will receive a second round of intratumoral injections into the same tumors selected for injections on day 1. Urine will also be collected right before the subject goes home.

STUDY VISIT 3:

The day 8 visit is identical to the day 4 visit. The same blood samples and urine sample are taken.

STUDY VISIT 4:

On the day 15 visit blood samples and a urine sample will be taken as well as a biopsy from one of the tumors.

Subjects will have to stay overnight at the hospital after each treatment.

FOLLOW UP:

A follow-up visit will be scheduled on days 29 where only blood samples and a urine sample will be taken.

The end of trial visit is scheduled around day 43 where in addition to lab samples a PET-CT scan will be performed.

Following day 43 the subject will be contacted by study staff at 6 week intervals for 3 months, then at 3 month intervals for up to one year and yearly thereafter.

ELIGIBILITY:
INCLUSION CRITERIA:

1. Age 18 - 70 years
2. Histologically-confirmed, advanced/metastatic solid tumor that is relapsed and/or refractory to standard therapy (progressive disease despite therapy).
3. Cancer is not surgically resectable for cure.
4. At least one measurable tumor mass by PETCT (i.e. PET-positive lesion that can reliable be assessed for SUV (standard update value) peak/SUV max, typically featuring longest diameter greater than or equal to 1 cm) and that can be injected by direct visualization/palpitation or by imaging-guidance (ultrasound)
5. Tumor suitable for biopsy. Biopsy is to be performed twice during the study (day 1 and day 15). The aim is to biopsy the same tumor at these visits.
6. Expected survival for approximately 12 weeks or longer
7. Performance Status WHO (World Health Organization) 0-2
8. Total bilirubin less than or equal to ULN (Upper Limit of Normal)
9. AST (Aspartate transaminase), ALT (Alanine aminotransferase) less than or equal to 3.0 × ULN
10. Serum creatinine less than or equal to 1.5 x ULN
11. INR (International Normalized Ratio) less than or equal to 1.5 x ULN
12. Hematologic parameters: Patients can be transfused to meet these entry criteria:

    1. Hemoglobin greater than or equal to 10 g/dL
    2. Leucocytes greater than or equal to 2300/mL
    3. platelet count greater than or equal to 75,000 plts/mm
13. Willing to participate as demonstrated by signed informed consent form.

EXCLUSION CRITERIA:

1. Known brain metastases or glioma. Central Nervous System malignancy, including carcinomatosis meningitis.
2. Tumor in the immediate pericardial vicinity
3. Use of high dose systemic corticosteroids or other immune suppressive medication within 3 weeks of first treatment.

   Note: patients taking low-dose corticosteroids for the treatment of nausea and/or taking maintenance corticosteroids for adrenal insufficiency are permitted to enroll.
4. Known infection with HIV (Human immunodeficiency virus) as this would affect the immune response of treatment or known underlying genetic immunodeficiency disease
5. Treatment of the injected tumor(s) with radiotherapy, chemotherapy, surgery, or an investigational drug within 4 weeks prior to first treatment.
6. Use of anti-viral medication. [Patients who discontinue such medications within 7 days prior to first treatment may be eligible for this study.]
7. Recent thromboembolic event
8. Clinically significant active infection or uncontrolled medical condition considered high risk for investigational new drug treatment (e.g. pulmonary, neurological, cardiovascular, metabolic such as type 2 diabetes, clinically significant and/or rapidly accumulating ascites, peri-cardial and/or pleural effusions)
9. Severe or unstable cardiac disease.
10. Current, active, progressing CNS (Central nervous system) malignancy, including carcinomatosis meningitis (definitively surgically resected or irradiated metastases allowed)
11. Pulse oximetry O2 (oxygen) criterion <90% at rest on room air
12. Vaccination with a live virus (i.e. measles, mumps, rubella, etc) < 30 days prior to first treatment
13. History of hepatic dysfunction, cirrhosis, hepatitis or malaria
14. Evidence of coagulation disorder
15. Women who are pregnant or nursing an infant
16. Previous organ transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Safety of CGTC-102 in patients with solid tumors | 28 days
  To assess the safety of the maximum tolerated dose and/or maximum feasible dose of CGTG-102 administered by intratumoral injection in a patient population with unresectable, refractory solid tumors
Efficacy of CGTC-102 in patients with solid tumors | 28 days
  To determine the maximum tolerated dose and/or maximum feasible dose of CGTG-102 administered by intratumoral injection in a patient population with unresectable, refractory solid tumors

SECONDARY OUTCOMES:
Development of tumor following the injection | 43 days
  To measure the development of adenovirus and tumor specific humoral responses following virus injection
Development of cellular immune response following the injection | 43 days
  To measure the development of cellular immune responses following virus injection

CONTACTS AND LOCATIONS:
Overall Officials: Martha M Pritchett, MD, Principal Investigator — Baylor College of Medicine